CLINICAL TRIAL: NCT04818892
Title: Immunogenicity of COVID-19 Vaccine in Patients With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0043; A534250 (Other: UW Madison); SMPH/MEDICINE/GASTROENT (Other: UW Madison); Protocol Version 6/6/2022 (Other: UW Madison); MSN252947 (Other Grant/Funding Number: AMERICAN COLLEGE OF GASTROENTEROLOGY); MSN253788 (Other Grant/Funding Number: TAKEDA PHARMACEUTICALS USA INC)
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: IBD; Covid19 Vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples for IBD specific research
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD and Non-Immunosuppressive Group: Clinical diagnosis of IBD, non-systemic immunosuppressive therapies, and scheduled to take an mRNA vaccine for COVID-19
  Interventions: Diagnostic Test: Serological Assay for SARS-CoV-2
- IBD and Immunosuppressive Group: Clinical diagnosis of IBD, treated with systemic immunosuppressive therapies, and scheduled to take an mRNA vaccine for COVID-19
  Interventions: Diagnostic Test: Serological Assay for SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: Serological Assay for SARS-CoV-2 — LabCorp's Cov2Quant IgG™ assay which uses immunoassay that uses electrochemiluminescent technology (ECL) for quantitative determination of anti-receptor binding domain (RBD) IgG antibodies specific to SARS-CoV-2.

SUMMARY:
The overall objective of this proposal is to evaluate the safety and immunogenicity of a COVID-19 vaccine in patients with Inflammatory Bowel Disease (IBD). This will help determine if immunosuppressive regimens impact COVID-19 vaccine response. The investigators will determine if certain groups may need more doses of a vaccine, with future adjuvanted vaccines or require a booster to maintain immunity. 260 participants with IBD and scheduled to get a COVID-19 vaccine will be recruited and can expect to be on study for 18 months.

DETAILED DESCRIPTION:
COVID-19 has a variable spectrum of illness with the majority of infection resulting in asymptomatic or mild disease. However certain healthy adults and immunosuppressed populations can develop severe or critical symptoms that require hospitalization or intensive care stay. Emerging evidence suggest that certain immunosuppressive medications used to treat patients with IBD such as anti-tumor necrosis factor (TNF) do not appear to confer an increased risk for severe COVID-19, but the risk appears to be higher for other agents such as corticosteroids. The efficacy of a candidate COVID-19 may be lower in immunosuppressed patients with IBD, since these patient populations may have lower responses to vaccines. Multiple studies have shown that patients with IBD have variability in their vaccine responses compared to healthy individuals. While many patients have a normal vaccine response, those treated with TNF agents or combination therapy (TNF inhibitors and immunomodulators) are more likely to mount a poor immune response. Furthermore, preliminary data suggest some novel regimens (such as vedolizumab) may not impact the immune response but there is insufficient data to know their impact on vaccine response. Thus, there is a critical need to determine whether patients with IBD will mount normal immune responses to a COVID-19 vaccine.

This is a single center cross sectional clinical study of 260 patients with IBD who are receiving the COVID-19 vaccine as standard of care. After obtaining informed consent, individuals who meet the inclusion criteria and none of the exclusion criteria will be invited to participate in the study.

Aim 1. Determine the immunogenicity and safety of a COVID-19 vaccine in patients with IBD. To achieve this aim, the investigators will perform a prospective study evaluating the immunogenicity of a COVID-19 vaccine in 260 patients with IBD.

* Hypothesis: Systemic immunosuppressive regimens such as Anti-TNF in combination with an immunomodulator, associated with the lowest vaccine response, or other systemic immunosuppressive regimens will blunt the immunogenicity of a COVID-19 vaccine while other agents such as vedolizumab or aminosalicylates will not affect the vaccine response.

Aim 2. Determine the impact of systemic immunosuppression on sustained antibody COVID-19 concentrations in patients with IBD who received the COVID-19 vaccine. To achieve this aim, the investigators will evaluate sustained antibody concentrations using a quantitative assay from LabCorp that is currently being used by the Centers for Disease Control and Prevention (CDC) to evaluate seroprevalence and study immunity at 1, 6, 12, and 18 months after completion of vaccination. Labcorp activities are provided as a fee for service. Follow up In-Person visit 1 (one month visit) will be optional and participants can enter the study at the six months study visit (Follow up In-Person visit 2) or at approximately 1-2 month post third dose of the COVID-19 vaccine which has been approved for patients with IBD. The 12 month visit (Follow up In-Person visit 3) may be replaced by a 6 month post 3rd dose vaccine if participants received one booster, or1-2 months post a 4th dose vaccine if participants received a second booster. The 18 month visit (Follow up In-Person visit 4) may substitute for a 12, 6, or 1-2 months post vaccine, depending on when and how many boosters the participant received.

* Hypothesis: Vaccine-induced antibody concentrations will wane over the 12 month interval faster than the published rate in healthcare workers.

At the completion of the proposed research, the safety and immunogenicity of a COVID-19 vaccine in immunosuppressed patients with IBD will be determined.

Protocol Amendment Approved 2/24/2022 changes time points of data collection to 18 months post-2nd dose, 9 month post-3rd dose, or 3-4 months post-4th dose.

Protocol Amendment Approved 4/19/2022 changes time points of data collection to 18 months post-2nd dose, 12 month post-3rd dose, or 6 months post-4th dose.

Protocol Amendment Approved 6/21/2022 indicates that follow up In-Person Visit 4 (will occur from July-October 2022 prior to a Fall 2022 COVID-19 booster. This blood draw can occur at any time after completion of any doses of a COVID-19 vaccine series). For participants who have not completed Visit 3 prior to July 2022, Visit 3 will be their last blood draw, which can occur from July-October 2022 prior to a Fall 2022 COVID-19 booster. This blood draw can occur at any time after completion of any doses of a COVID-19 vaccine series).

ELIGIBILITY:
Inclusion Criteria:

For mRNA cohort:

* Participant has a history of ulcerative colitis (UC) or Crohn's disease diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria.
* On one of the following treatment regimens:

  * Group A: Non-systemic immunosuppressive Group at least 75 participants

    * Mesalamine monotherapy or no therapy for IBD
    * Vedolizumab Therapy Group: on either vedolizumab monotherapy or combination therapy with methotrexate or azathioprine
  * Group B: Systemic immunosuppressive Group at least 75 participants

    * Thiopurine Therapy Group: on azathioprine at least 2.0mg/kg or 6MP 1.0mg/kg
    * Anti-TNF Therapy Group: on maintenance therapy infliximab (at least 8 every 8 weeks), golimumab (at least monthly), adalimumab (at least every 2 weeks), or certolizumab (at least monthly)
    * Anti-TNF Combination Therapy Group: on anti-TNF therapy as described above along with either 15mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg
    * Ustekinumab Therapy Group: on either ustekinumab monotherapy or combination therapy with methotrexate or azathioprine.
    * Tofacitinib Therapy Group: on tofacitinib at least 5mg PO BID
    * Corticosteroid Therapy Group: on any one of the systemic immunosuppressive groups and any dose of corticosteroids
* Participant has been on the same IBD treatment for at least two months.
* Participant is receiving an mRNA COVID-19 vaccine per standard of care recommended by their clinical provider or has started the COVID-19 series or finished the mRNA COVID-19 vaccine series within the past six months and would qualify for six month study visits or has received a third dose of the vaccine as standard of care.
* Participants entering in the study at the six month study visit must have been on same treatment at their time of immunization.

For Viral vector cohort:

* Participant has a history of ulcerative colitis (UC) or Crohn's disease diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria.
* On one of the following treatment regimens:

  * Group A: Non-systemic immunosuppressive Group at least 15 participants

    * Mesalamine monotherapy or no therapy for IBD
    * Vedolizumab Therapy Group: on vedolizumab monotherapy
  * Group B: Systemic immunosuppressive Group at least 15 participants

    * Thiopurine Therapy Group: on azathioprine at least 2.0mg/kg or 6MP 1.0mg/kg
    * Anti-TNF Therapy Group: on maintenance therapy infliximab (at least 8 every 8 weeks), golimumab (at least monthly), adalimumab (at least every 2 weeks), or certolizumab (at least monthly)
    * Anti-TNF Combination Therapy Group: on anti-TNF therapy as described above along with either 15mg of methotrexate or azathioprine at least 1.0mg/kg or 6MP 0.5mg/kg
    * Ustekinumab Therapy Group: on either ustekinumab monotherapy or combination therapy with methotrexate or azathioprine.
    * Tofacitinib Therapy Group: on tofacitinib at least 5mg PO BID
    * Corticosteroid Therapy Group: on any one of the systemic immunosuppressive groups and any dose of corticosteroids
* Participant has been on the same IBD treatment for at least two months.
* Participant is receiving a viral vector COVID-19 vaccine per standard of care or has started or finished the viral vector series within the past 6 months. If participant entering at six months and would qualify for six month study visits and has received an additional one or two dose of viral vector of mRNA for a total of two -three COVID vaccines as standard of care.
* Participants entering in the study at the six month study visit must have been on same treatment at their time of immunization.

Exclusion Criteria:

For mRNA cohort:

* Allergy to COVID-19 vaccine or a component of it
* Participant cannot or will not provide written informed consent
* Unable to provide appropriate informed consent due to being illiterate or impairment in decision-making capacity

For Viral vector cohort:

* Allergy to COVID-19 vaccine or a component of it
* Participant cannot or will not provide written informed consent.
* Unable to provide appropriate informed consent due to being illiterate or impairment in decision-making capacity.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with IBD and scheduled to receive a COVID-19 vaccine will be recruited from the University of Wisconsin Hospital and Clinics if they meet the inclusion and exclusion criteria.
  * Group A IBD patients on non-systemic immunosuppressive therapy: no therapy or aminosalicylates or vedolizumab therapy
  * Group B IBD patients on systemic immunosuppression
  Patients in both groups will have been on stable treatment for IBD for at least two months.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Change in Geometric Mean Titers (GMT) of SARS-CoV-2 Antibody Concentrations following mRNA COVID-19 vaccine series | baseline to 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  The primary endpoint will be evaluating the change in humoral immunity between the immunosuppressive and non-immunosuppressive IBD treatment regimens following the recommended doses mRNA COVID-19 vaccine series.
Sustained antibody concentrations of mRNA COVID-19 vaccines | 18 months post-2nd dose
  The investigators will evaluate sustained antibody concentrations of mRNA COVID-19 vaccines by using a quantitative assay from LabCorp that is currently being used by the CDC to evaluate seroprevalence.
Sustained antibody concentrations of mRNA COVID-19 vaccines | 12 months post-3rd dose
  The investigators will evaluate sustained antibody concentrations of mRNA COVID-19 vaccines by using a quantitative assay from LabCorp that is currently being used by the CDC to evaluate seroprevalence.
Sustained antibody concentrations of mRNA COVID-19 vaccines | 6 months post-4th dose
  The investigators will evaluate sustained antibody concentrations of mRNA COVID-19 vaccines by using a quantitative assay from LabCorp that is currently being used by the CDC to evaluate seroprevalence.
Change in level of T-cell response after mRNA COVID-19 vaccine | 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  Investigators will evaluate sustained cell mediated immunity against Covid-spike proteins after completing the vaccine schedule of a mRNA COVID-19 vaccine.
Percentage of participants with detectable level of T-cell response after mRNA COVID-19 vaccine | 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  For each patient, peripheral blood monocytes (PBMCs) will be isolated. IFN-ϒ ELISpot, which detects both CD4 and CD8 T cell effectors, will be used to detect T-cell immunity to the Covid-spike protein or peptides. The plates will be read on an AID ELISpot reader (Cell Technology, Inc., Columbia MD, reader software v.3.1.1.). A positive response to antigen will be defined as a frequency that was significantly (p < 0.05, two-tailed t test) greater than the mean of control no-antigen wells and detectable (i.e., >1:100,000). T cell responses will be correlated to Covid-19 neutralizing antibody responses.

SECONDARY OUTCOMES:
Incidence of Adverse Events | up to 1 month post final immunization
  Safety will be assessed by the incidence of adverse events (AEs and SAEs) related to the vaccine.
Patient reported outcome 3 (PRO3) score | baseline, 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  Safety will be assessed by monitoring the PRO3 scores at baseline and 1 month post-vaccination. PRO-3 is a measure of overall well-being as well as specific symptoms and complications of CD, such as stool frequency, abdominal pain and general well being. Greater PRO3 scores indicate more severe CD symptoms.
Simple Colitis Activity Index (SCAI) Questionnaire Score | baseline, 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  For participants with Ulcerative Colitis (UC), safety will be assessed by monitoring the SCAI score at baseline and 1 month post-vaccination. SCAI is a measure of overall well-being as well as specific symptoms and complications of UC, such as stool frequency and abdominal pain. The total possible range of scores is 0-21, with higher scores indicative of increased symptoms.
Seroconversion: assessed by percentages of participants with ≥4-fold rise in antibody titer | 1 month post-immunization
  Percentages (and 2-sided 95% CIs) of participants with ≥4-fold rise will be assessed for the COVID-19 vaccine within each group.
Change in Geometric Mean Titers (GMT) of SARS-CoV-2 Antibody Concentrations following two doses of viral vector COVID-19 vaccine series | baseline,18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  The primary endpoint will be evaluating the change in humoral immunity between the immunosuppressive and non-immunosuppressive IBD treatment regimens following the two doses viral vector COVID-19 vaccine series.
Sustained antibody concentration of viral vector COVID-19 vaccines | 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  The investigators will evaluate sustained antibody concentrations of viral vector COVID-19 vaccines by using a quantitative assay from LabCorp that is currently being used by the CDC to evaluate seroprevalence.
Percentage of participants with detectable level of T-cell response after viral vector COVID-19 vaccine | 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  For each patient, peripheral blood monocytes (PBMCs) will be isolated. IFN-ϒ ELISpot, which detects both CD4 and CD8 T cell effectors, will be used to detect T-cell immunity to the Covid-spike protein or peptides. The plates will be read on an AID ELISpot reader (Cell Technology, Inc., Columbia MD, reader software v.3.1.1.). A positive response to antigen will be defined as a frequency that was significantly (p < 0.05, two-tailed t test) greater than the mean of control no-antigen wells and detectable (i.e., >1:100,000). T cell responses will be correlated to Covid-19 neutralizing antibody responses.
Change in level of T-cell response after viral vector COVID-19 vaccine | 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  Investigators will evaluate sustained cell mediated immunity against Covid-spike protein after completing the vaccine schedule of a viral vectors vaccine.
Presence of SARS-CoV2 anti-nucleocapside antibody : Yes/No | baseline, 18 months post-2nd dose, 12 months post-3rd dose, or 6 months post-4th dose
  To evaluate the rate of asymptomatic COVID-19 infections in patients with IBD, investigators will evaluate the presence for anti-nucleocapside antibody in participants at baseline and/or 1 month visit after immunization to evaluate the rate of asymptomatic infection in our cohort. A SARS-CoV2 anti-nucleocapside antibody is not induced by vaccine so it's presence means there was a presence of a previous infection.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Caldera, DO, MS, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No